CLINICAL TRIAL: NCT03205254
Title: Short-term Effects of Mediterranean or Fast Food Diet on HDL Composition and Function
Brief Title: Effects of Short-term Diet on HDL Composition and Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 801116; UCDAMZ2 (Other: UC Davis)
Record Dates: First submitted 2017-06-27; First posted 2017-07-02 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Diet Modification; HDL; Inflammation
Keywords: Mediterranean diet; HDL; Fast food; Gut microbiota; Inflammation
MeSH Terms: conditions — Inflammation | interventions — Diet, Mediterranean

STUDY DESIGN:
Intervention Model Description: Randomized two-way crossover design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Active Comparator): Participants randomized to group A follow the 4-day Mediterranean diet and then the 4-day fast food diet with a 4-day washout period in between.
  Interventions: Other: Mediterranean Diet; Other: Fast food diet
- Group B (Active Comparator): Participants randomized to group B follow the 4-day fast food diet and then the 4-day Mediterranean diet with a 4-day washout period in between.
  Interventions: Other: Mediterranean Diet; Other: Fast food diet

INTERVENTIONS:
Other: Mediterranean Diet — four days of participant-scaled isocaloric Mediterranean meals
Other: Fast food diet — four days of participant-scaled isocaloric fast food meals

SUMMARY:
The primary objective of this study is to generate preliminary data on the effects of a short-term diet of either fast food or Mediterranean type diet on HDL and microbiota composition and function in healthy subjects, which includes both normal weight and overweight/obese subjects.

DETAILED DESCRIPTION:
Subjects will be recruited through word-of-mouth, flyers, newspaper advertisements, and postings on the UC Davis Nutrition Department website. Interested individuals who respond to notices will undergo a telephone screen to assess eligibility. A copy of the flyer, the Nutrition Department website notice, newspaper advertisement, and phone screen are attached with this submission. The subject population may reflect the ethnic and cultural diversity of the region.

Screening and Consent Prospective subjects who pass the initial phone screening interview (i.e. meet inclusion/exclusion criteria) will be admitted into the study and scheduled for a consent visit. At the consent visit, after singing the consent form and agreeing to participate, participants' weight, height, and blood pressure will be measured to ensure that they meet inclusion criteria, and if their measurements agree with their reported values they will be admitted into the study and scheduled for their baseline visit. At the consent visit, subjects will also be instructed on how to complete a 3-day food record and will be asked to complete and return it before the baseline visit. Participants will also be given a stool collection kit during the consent visit to collect stool samples within 24 hours before their first scheduled visit. Women who consent to participate will be scheduled to complete the study within the luteal phase and menses of the menstrual cycle to avoid confounding alterations in lipoproteins. If women participants are not able to remember the first day of their last menstrual cycle, they will be instructed to note the start of their next menstrual cycle and will then be scheduled accordingly thereafter. Subjects will be randomized to begin either on the fast food arm or the Med arm. Each cohort of 4 participants will have 2 individuals who begin on the Med diet arm, and 2 individuals who begin on the fast food diet arm, and each participant will be randomized into one of these two blocks and be assigned a study ID number.

Baseline Visit A At the scheduled baseline visit subjects will report to the Ragle Human Nutrition Research Center located on the UC Davis campus (1283 Academic Surge, University of California, Davis, in Davis CA 95616) for a 12-hour fasting blood draw and anthropometric measurements. They will be asked to bring their stool sample to this visit. Each participant will also be asked to complete a health history questionnaire, a physical activity questionnaire, and a Food Frequency Questionnaire (FFQ). The duration of the baseline study visit will be approximately 1 hour.

Study Arm 1: (4 days) Following the baseline blood draw, subjects randomized to begin on the fast food arm will consume a fast food diet for 4 days, Subjects randomized to begin on the Med diet arm will consume foods provided to them and follow basic food preparation instructions. At the end of each 4-day-long diet phase, subjects will report to the Ragle Human Nutrition Research Center again for their first follow-up study visit (Study Visit 2). Participants will be required to collect another stool sample to bring with them to their visit and will complete a hunger and satiety questionnaire at either the lunch or dinner meal each day on each diet arm.

During the Med diet arm, participants will pick up their meals and instructions from the study team. During the fast food diet arm, participants will be given gift cards and meal plans to follow for the on-campus fast food restaurants and will purchase meals at the fast food restaurants on their own. For both dietary interventions, participants will follow the appropriate meal plan, attached with this submission. They will also be instructed to maintain their physical activity level during the study period. Subjects will be contacted once during each dietary period by e-mail or phone and will be asked about their general wellbeing, and to remind them to collect a stool sample for the next visit. To monitor compliance, participants will fill out a compliance survey as well as bring in any leftover food they do not consume. The leftover foods plus packaging will be weighed, and the weight of packaging alone subtracted in order to obtain an accurate measurement of how much participants actually consumed.

Study Visit B This study visit will also be approximately 1 hour in duration, and will also include a fasting blood draw, anthropometric measurements, and the same questionnaires as the baseline study visit except they will not complete an FFQ. Participants will receive the first installment of their study compensation at this time.

Study Washout Period: (4 days) Following Study Visit B, subjects will enter a 4-day washout period, in which they will return to their normal diets. Subjects will be required to complete a 3-day food record during this time. At the end of the 4-day washout period, subjects will return to the Ragle facility for the second follow-up Visit (Study Visit C). Participants will be required to collect another stool sample to bring with them to their visit.

Study Visit C This study visit will also be approximately 1 hour in duration, and will also include a fasting blood draw, anthropometric measurements, and the same questionnaires as study visit B. Participants will receive the second installment of their study compensation at this time.

Study Arm 2: (4 days) At this time, participants who completed the mMed diet arm will now begin the fast food diet arm, and those who completed the fast food diet arm will now enter the mMed diet arm. All participants will be asked to complete a hunger and satiety questionnaire during this time (4 days). At the end of the 4-day period subjects will return for the third follow-up study visit (Study Visit D). Participants will be required to collect a final stool sample to bring with them to their visit.

Study Visit D This study visit will also be approximately 1 hour in duration, and will also include a fasting blood draw, anthropometric measurements, and the same questionnaires as study visits B and C. Subjects will receive the rest of their compensation at this time.

ELIGIBILITY:
Inclusion Criteria:

* 19-30 years old (women and men)
* Weigh 133 pounds (60.5kg) or more
* Currently consuming fast food 4 times per week or less
* Categorized in "any" of the following BMI ranges:

  1. BMI: 18.5-25 kg/m², for the group of healthy subjects with optimal body weight
  2. BMI: 26-35 kg/m², for the group of overweight/obese subjects
* Willing to consume a healthy diet (i.e. low saturated fat, low refined carbohydrate, high fruit and vegetable, high fiber) for 4 days.
* Willing to consume a fast food diet (i.e. high saturated fat, high refined carbohydrate, low fruit and vegetable, low fiber) for 4 days, including a beef burger twice a day
* Willing to bring all unfinished food (except beverages) back to Ragle facility in a plastic Ziploc bag.
* Willing to bring in receipts from fast food purchases

Exclusion Criteria:

* Smoker
* Anemia
* Food allergies
* Intolerance to dairy or gluten
* Pregnant or lactating
* Irregular menstrual cycle
* Change in hormonal contraceptive use within the previous 3 months
* Documented chronic diseases including diabetes, thyroid disease, metabolic syndrome, cancer (active), or previous cardiovascular events
* Current consumption more than 1 alcoholic drink/day
* Current consumption of fast food more than 4 times per week
* Fish consumption greater than or equal to 3 times per week
* Extreme dietary or exercise patterns
* Recent weight fluctuations (greater than 10% in the last six months)
* Taking prescription lipid medications (e.g. statins) or other supplements known to alter lipoprotein metabolism such as isoflavones.
* Visit 1 baseline glucose: >100 mg/dL
* Regular use (> 1 time per week) of allergy or pain medications

Ages: 19 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-03-28 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
HDL ApoA-I content | 24 months
  Measure the concentration of ApoA-I in isolated HDL by ELISA

SECONDARY OUTCOMES:
HDL lipidomic composition | 24 months
  Measure lipidomic composition of isolated HDL by LC-MS
HDL proteomic composition | 24 months
  Measure proteomic composition of isolated HDL by LC-MS
HDL cholesterol efflux capacity | 24 months
  Measure capacity of isolated HDL to efflux cholesterol out of macrophages
HDL anti-inflammatory capacity | 24 months
  Measure capacity of isolated HDL to modify cytokine secretion in macrophages
Gut microbiome changes | 24 months
  Measure gut microbiota composition by 16S sequencing of stool samples

CONTACTS AND LOCATIONS:
Overall Officials: Angela Zivkovic, PhD, Principal Investigator — UC Davis Nutrition Department
Locations (1):
- UC Davis Ragle Center for Human Nutrition, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhu C, Sawrey-Kubicek L, Beals E, Rhodes CH, Houts HE, Sacchi R, Zivkovic AM. Human gut microbiome composition and tryptophan metabolites were changed differently by fast food and Mediterranean diet in 4 days: a pilot study. Nutr Res. 2020 May;77:62-72. doi: 10.1016/j.nutres.2020.03.005. Epub 2020 Mar 26. PMID 32330749
- [Result] Zhu C, Wong M, Li Q, Sawrey-Kubicek L, Beals E, Rhodes CH, Sacchi R, Lebrilla CB, Zivkovic AM. Site-Specific Glycoprofiles of HDL-Associated ApoE are Correlated with HDL Functional Capacity and Unaffected by Short-Term Diet. J Proteome Res. 2019 Nov 1;18(11):3977-3984. doi: 10.1021/acs.jproteome.9b00450. Epub 2019 Oct 1. PMID 31545048
- [Result] Zhu C, Sawrey-Kubicek L, Beals E, Hughes RL, Rhodes CH, Sacchi R, Zivkovic AM. The HDL lipidome is widely remodeled by fast food versus Mediterranean diet in 4 days. Metabolomics. 2019 Aug 17;15(8):114. doi: 10.1007/s11306-019-1579-1. PMID 31422486